CLINICAL TRIAL: NCT00750958
Title: PREVENT - Prospective Rhythm Event Surveillance in the ER With NetGuard
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Datascope Patient Monitoring (Industry)
Responsible Party: Dr. Charles Pollack, Jr., Pennsylvania Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 807119
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Cardiac Event
Keywords: cardiac rhythm changes
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (No Intervention): ED patients that are not monitored with conventional therapy.
  Interventions: Procedure: NetGuard Automated Clinician Alert System

INTERVENTIONS:
Procedure: NetGuard Automated Clinician Alert System — Monitoring System for in-hospital patients who are typically unmonitored. Identifies and alarms for cardiac rhythm changes.
  Other Names: NetGurard Automated Clinican Alert Systemm

SUMMARY:
The purpose of this study is to determine the incidence of clinically significant rhythm and rate changes in ED patients who are not placed on conventional telemetry, and to test the user-friendliness of a automated clinician alter device in hectic and noisy setting of a busy emergency room.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yes
* Agree to participate in study
* Telemetry not indicated
* Telemetry not available
* Willingness to complete a questionnaire-

Exclusion Criteria:

* Refusal to participate
* Know sensitivity to adhesive
* Language/communication barriers
* Perceived high risk for lack of study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant rhythm and rate changes in ED patients. | Patient ED stay

SECONDARY OUTCOMES:
Measure of user-friendliness of the device. | Patient ED stay

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pollack, MD, Principal Investigator — Pennslvania Hospital
Locations (2):
- United States (2):
  - Dr Charles Pollack, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania